CLINICAL TRIAL: NCT07216391
Title: Adaptive Platform Trial to Delay Progression From Stage 2 to Stage 3 Type 1 Diabetes: Comparing Teplizumab With Low-dose Anti-Thymocyte Globulin (ATG) Protocol TN-40A
Brief Title: Platform Trial to Delay Stage 3 Diabetes: Comparing Teplizumab With ATG
Acronym: TN40A
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TN40A
Record Dates: First submitted 2025-09-22; First posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: TrialNet; T1D; Teplizumab; ATG
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Antilymphocyte Serum; teplizumab

STUDY DESIGN:
Intervention Model Description: This trial will enroll 60 participants who will be randomly assigned in a 2:1 allocation to the following treatment arms: 40 participants will be randomized to ATG and 20 participants will be randomized to teplizumab.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ATG (Experimental): Antithymocyte globulin (ATG) will be intravenously administered over two days, with a total of 2 infusion periods. The first dose (0.5mg/kg) will be infused over a minimum of 6 hours, and the second dose (2mg/kg) over a minimum of 4 hours with a maximum infusion time for each infusion of 10 hours. Infusions may be administered either in a hospital or outpatient setting at the investigator's or institutions discretion.
  Interventions: Drug: Antithymocyte Globulin (ATG)
- Teplizumab (Active Comparator): Intravenous infusions of teplizumab will be given for 14 consecutive days. Each infusion takes about 30 minutes. Vital signs will be monitoring for at least 30 minutes after each infusion. If reactions to the infusion occur participants may be monitored for at least 2 hours after the study drug infusion. The total dose for the 14-day course is approximately 11,240 µg/m².
  Interventions: Drug: Teplizumab

INTERVENTIONS:
Drug: Antithymocyte Globulin (ATG) — Thymoglobulin
  Arms: ATG
Drug: Teplizumab — Intravenous infusions of teplizumab given for 14 consecutive days. Each infusion takes about 30 minutes and is followed by an observation period of at least 30 minutes.
  Arms: Teplizumab

SUMMARY:
This is a 2-arm, multi-center, open label study to learn if ATG works the same or better than teplizumab in delaying or preventing Stage 3 Type 1 diabetes. Participants will be administered either 2 infusions of ATG or 14 infusions of teplizumab and will be followed for 12 months after administration.

DETAILED DESCRIPTION:
This protocol will enroll 60 participants with Stage 2 diabetes. Oral glucose tolerance testing will be done at the screening, baseline visit (V0) and at 3, 6 and 12 months after study drug administration. Participants will continue follow-up visits until 12 months from the baseline visit.

ELIGIBILITY:
Inclusion Criteria:

* Willing to provide informed consent or have a parent or legal guardians provide informed consent when the participant is <18 years of age.
* Aged ≥4 to <35 years
* A history of at least two or more diabetes-related biochemical autoantibodies (mIAA, GADA, ICA, IA-2A, ZnT8A) present on the same sample. In the absence of other antibodies, ICA and GADA positivity alone will not suffice for eligibility in this trial.
* Participants must meet ADA stage 2 T1D glycemic criteria* by TrialNet testing within 100 days of randomization.

  *The ADA definition of stage 2 T1D is characterized by glucose intolerance or dysglycemia in the presence of two or more islet autoantibodies, impaired fasting glucose (≥ 100mg/dL), impaired glucose tolerance (2-hour post 75g glucose load ≥ 140mg/dL), high glucose levels at intermediate time points on OGTT (30, 60, 90 min timepoints of ≥ 200 mg/dL), and/or HbA1c between 5.7% and 6.4% or ≥ 10% increase in HbA1c within a two year window, with the most recent HbA1c value obtained within 100 days of randomization.
* CMV and/or EBV seronegative participants must be CMV and EBV PCR negative within 30 days of randomization and may not have had signs or symptoms of a CMV or EBV-compatible illness lasting longer than 7 days within 30 days of randomization.
* CMV seropositive participants must be CMV PCR negative and all EBV seropositive participants must have EBV PCR < 2,000 IU/mL within 30 days of randomization and may not have had signs or symptoms of a CMV or EBV-compatible illness lasting longer than 7 days within 30 days of randomization.
* Be at least 4 weeks from last live immunization.
* Be willing to forgo vaccines (other than non-live influenza and COVID-19) during the 3 months after study drug treatment period.
* Must meet TrialNet eligibility minimum immunization recommendations found in Appendix A of the manual of operations (MOO).
* With the exception of stage 2 T1D, participants must be healthy, as defined by absence of any other untreated diagnoses that the investigator deems to be a potential confounder.
* If a female participant with reproductive potential, willing to avoid pregnancy (abstinence or adequate contraceptive method) through the completion of the study infusions and up to 3 months after study drug administration and undergo pregnancy testing prior to each study visit.
* Must be residing or have accommodations within 1 hour of the infusion site during study drug infusions and must be within 1 hour of a medical care facility for 1 day after completion of infusions.
* Participants must live in a location with rapid access to emergency medical services.

  * The ADA definition of stage 2 T1D is characterized by glucose intolerance or dysglycemia in the presence of two or more islet autoantibodies, impaired fasting glucose (≥ 100mg/dL), impaired glucose tolerance (2-hour post 75g glucose load ≥ 140mg/dL), high glucose levels at intermediate time points on OGTT (30, 60, 90 min timepoints of ≥ 200 mg/dL), and/or HbA1c between 5.7% and 6.4% or ≥ 10% increase in HbA1c within a two year window, with the most recent HbA1c value obtained within 100 days of randomization.

Exclusion Criteria:

* Immunodeficiency or clinically significant chronic lymphopenia: (Leukopenia (<3,000 leukocytes/μL), neutropenia (<1,500 neutrophils/μL), lymphopenia (<800 lymphocytes/μL), thrombocytopenia (<100,000 platelets/μL).
* Active signs or symptoms of acute or chronic infection at the time of randomization including SARS-Cov-2.
* Uncontrolled autoimmune thyroid disease and/or celiac disease (participants must be well controlled for the previous 6 months).
* Evidence of a history of prior or current tuberculosis infection as assessed interferon gamma release assay (QuantiFERON) with the exception of post-exposure prophylaxis.
* Currently pregnant or lactating or anticipate getting pregnant within the study period.
* Require use of other immunosuppressive agents including chronic use of oral or intravenous injectable steroids.
* Evidence of current or past HIV or Hepatitis B or current Hepatitis C infection.
* Any complicating medical issues or abnormal clinical laboratory results that may interfere with study conduct, or cause increased risk to include pre-existing cardiac disease, COPD, sickle cell disease, neurological disease, or blood count abnormalities.
* A history of malignancies other than of skin.
* Evidence of liver dysfunction with AST or ALT ≥ 2 times the upper limit of the reference range.
* Evidence of renal dysfunction with creatinine ≥ 1.5 times the upper limit of the reference range.
* Increased bilirubin ≥ 2 times (total) or ≥ 1.5 times (direct) the normal limit (Participants with documentation of Gilbert's Disease permitted).
* Vaccination with a live vaccine within the last 4 weeks or killed/inactivated vaccine within the last 2 weeks.
* Current or ongoing use of non-insulin pharmaceuticals that affect glycemic control within 14 days of screening.
* Prior treatment with Teplizumab or ATG (either in a previous clinical trial or clinically).
* Has previously participated in a clinical trial for diabetes prevention and received active study agent within 6 months of treatment.
* Known allergy to rabbits or rabbit derived products.
* Prior adverse reactions to heparin.
* Any condition that in the investigator's opinion may adversely affect study participation.
* Any screening/baseline laboratory result not otherwise stated out of normal reference range and/or medical history that may increase the risk of the participant's participation in this trial.
* Previously diagnosed with Stage 3 TID according to ADA criteria.

Ages: 4 Years to 34 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in DPTRS at six months | 6 months after completion of study drug administration
  DPTRS is calculated as DPTRS = (1.569 x log-BMI) - (0.056 x age) + (0.813 x glucose sum from 30 to 120 min /100) - (0.848 x C-peptide sum from 30 to 120 min/10) + (0.476 x log-fasting C-peptide), where the units are years for age, kg/m2 for BMI, mg/dl for glucose, ng/ml for C-peptide

SECONDARY OUTCOMES:
Progression to Stage 3 T1D | 6 months after study drug administration
  Elapsed time from study drug administration to the development of diabetes or time of last contact among those randomized
OGTT glucose AUC | 6 months after study drug administration
  Mean area under the stimulated glucose curve (AUC) over the 2-hour oral glucose tolerance test.
M120 score | 6 months after study drug administration
  This is an aggregated score from multiple measurements calculated as follows:
  M120 = 0.448×(sex) + 0.631×(IA-2A) - 0.0302×(age) + 0.0605×(BMI)
  + 1.380×(HbA1c) + 0.0265×(120 min glucose) - 0.191×(120 min C-peptide), where the units for BMI, age, glucose, C-peptide and HbA1c are, respectively, kg/m2, years, mg/dl, ng/ml and percentage units. Sex was assigned a score of 1 for male and 2 for female, and IA-2A status assigned 0 for absent and 1 for present. Glucose is converted from mmol/l to mg/dl by multiplying by 18; C-peptide is converted from nmol/l to ng/ml by dividing by 3.00; and HbA1c is converted from mmol/mol to percentage units by adding 23.5 and then dividing by 10.93.
Index 60 | 6 months after study drug administration
  This is an aggregated score from multiple measurements calculated as follows:
  Index60 = 0.3695×loge(fasting C-peptide) + 0.0165×(60 min glucose) - 0.3644×(60 min C-peptide), where the units for glucose and C-peptide are, respectively, mg/dl and ng/ml. Glucose is converted from mmol/l to mg/dl by multiplying by 18; C-peptide is converted from nmol/l to ng/ml by dividing by 3.00.
OGTT C-peptide AUC | 6 months after study drug administration
  Mean area under the stimulated C-peptide curve (AUC) over the 2-hour oral glucose tolerance test
HbA1c | 6 months after study drug administration
  Measured as a percentage of total hemoglobin

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be available at the NIDDK Central Repository
Supporting Information: Study Protocol, ICF
Time Frame: Final datasets will be available at the NIDDK Central Repository 12 months from the last participant's follow-up visit
Access Criteria: IPD can be requested through the NIDDK Central Repository once submitted.

REFERENCES:
- See also: Related Info — https://www.trialnet.org/